CLINICAL TRIAL: NCT05009966
Title: A Phase I Trial to Evaluate Safety, Tolerability, Pharmacokinetics, Immunogenicity and Initial Efficacy of SYSA1801 in the Treatment of CLDN 18.2 Positive Advanced Malignant Solid Tumor
Brief Title: Study of SYSA1801 in the Treatment of Claudin( CLDN) 18.2 Positive Advanced Malignant Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1801-CSP-001
Record Dates: First submitted 2021-08-03; First posted 2021-08-18 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-08

CONDITIONS: Advanced Solid Tumor; Gastric Cancer (GC); Gastroesophageal Junction (GEJ) Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms; Pancreatic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SYSA1801 for injection (Experimental): Stage I: Dose Escalation and dose expansion： Dose Escalation：SYSA1801 will be administered intravenously (IV) at different dose levels, including 0.5, 1, 2, 3, 4.5 and 6 mg/kg according to a modified 3+3 dose-escalation design. Accelerated dose titration design will be used for the first 2 dose levels (0.5 and 1 mg/kg), and then traditional 3+3 dose escalation design will be used for the following levels (2, 3, 4.5 and 6 mg/kg).
  Dose expansion: SYSA 1801 will be administered at up to dose levels which is equal or lower than MTD IV infusion. Each dose level contains no more than 12 subjects (including subjects in dose escalation) Stage II: Extension cohort This cohort will comprise subjects with Claudin 18.2 positive GC or GEJ adenocarcinoma, pancreatic cancer or other solid cancer with prior failure of, progression on, or intolerance to, standard therapy.
  The starting dose of SYSA1801 for expansion will be derived from the RP2D determined during Stage I
  Interventions: Drug: SYSA1801 for injection

INTERVENTIONS:
Drug: SYSA1801 for injection — SYSA1801 will be administered intravenously (IV) on Day 1 of every 21-day cycle. Individual subjects may continue study treatment until there is evidence of disease progression (clinical or radiologic) judged by Investigators, unacceptable toxicity or other reasons for treatment discontinuation.

SUMMARY:
This is an open-label, dose escalation, dose expansion and extension cohort phase 1 study to evaluate the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of SYSA1801

DETAILED DESCRIPTION:
This study includes two stages. The dose escalation and dose expansion part (Stage I) will determine the MTD and RP2D of SYSA1801 in subjects with advanced solid tumor for which there is no available standard likely to confer clinical benefit based on a modified 3+3 dose escalation design (an accelerated dose titration design followed by traditional 3+3 dose escalation design) The extension cohort (Stage II) will evaluate the preliminary efficacy and safety of SYSA1801 in subjects with Claudin 18.2 positive gastric cancer (GC), gastroesophageal junction (GEJ) cancer, pancreatic cancer, non-small cell lung cancer and other solid tumors who have relapsed and/or are refractory to approved therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects provide documented informed consent voluntarily;
2. Male or female subjects ≥ 18 years and ≤ 75 years;
3. Subjects with locally advanced unresectable or metastatic malignant solid tumors confirmed by histology and/or cytology and CLDN 18.2 positive expression in the tumor tissue confirmed by the central laboratory: dose-escalation phase defined as IHC ≥ 1+ by central laboratory IHC assay; dose-expansion phase and extension cohort studies defined as CLDN18.2 expression in ≥ 40% of tumor cells, the IHC ≥ 2+);
4. Subjects met following requirements according to the different stages: Stage I: subjects have no standard treatment, or the standard treatment failed or was intolerant, or have no condition to receive standard treatment; Stage II: Subjects had received at least one prior line of systemic chemotherapy with clear disease progression confirmed by investigator or documented by medical records, in the following phase II cohorts:

   Cohort A: Gastric cancer/adenocarcinoma of gastroesophageal junction Cohort B: Pancreatic cancer Cohort C: Non-small cell lung cancer Cohort D: Other solid tumors expressing CLDN 18.2;
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0 or 1, and life expectancy ≥ 3 months;
6. At least one measurable lesion according to RECIST1.1;
7. The main organ function met the following criteria within 7 days before enrollment (no blood transfusion, EPO, G-CSF or other medical support treatment within 14 days before administration of study drug): neutrophil ≥ 1.5 × 10^9 /L, platelet ≥ 100 × 109/L, hemoglobin ≥ 90 g/L or ≥ 5.6 mmol/L; International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × Upper limit of normal range (ULN), activated partial thrombin time (APTT) ≤ 1.5 × ULN, serum creatinine ≤ 1.5 × ULN, total bilirubin (TBIL) ≤ 1.5 × ULN (≤ 3 × ULN for subjects with Gilbert's syndrome or liver metastasis), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for subjects with liver metastasis);
8. Fertile women must have negative pregnancy tests before study entry;
9. Men and fertile women must agree to take effective contraceptive measures from signing informed consent to 6 months after the last administration;
10. Understand the trial requirements, and willing to follow the trial and follow-up procedures.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Subjects who have not recovered from the adverse reactions caused by previous anti-tumor treatment (refer to NCI CTCAE 5.0, ≤ grade 1 or at baseline), except for the toxicity of alopecia, pigmentation and other conditions have no safety risk according to investigators' opinion;
3. Antitumor therapy such as chemotherapy, radiotherapy, biotherapy, targeted therapy, immunotherapy and other anti-tumor treatment within 4 weeks before administration of the study drug, and the following items: Nitrosourea (such as carmustine, lomustine, etc.) or mitomycin C were within 6 weeks before administration of the study drug; Oral fluorouracil and small molecule targeted drugs within 5 half-lives before administration of the study drug; Endocrine therapy or traditional Chinese medicines with anti-tumor indications within 2 weeks before administration of the study drug; Palliative radiotherapy for bone metastasis or local radiotherapy for pain relief within 2 weeks before administration of the study drug; Drugs for bone metastasis related events (such as zoledronic acid, etc.) did not affect the enrollment;
4. Subjects who have undergone major surgery (excluding needle biopsy) within 4 weeks before administration of the study drug, or who are expected to undergo major surgery during the study period, or who have severe unhealed wounds, trauma, ulcers, etc;
5. Subjects with previous intolerance to CLDN 18.2 monoclonal antibody or known components of SYSA1801, or severe allergic reactions;
6. Subjects with symptoms of brain or pia mater metastasis; Subjects with central nervous system (CNS) metastases in the following conditions can be considered: subjects with brain metastases without treatment and without symptoms, or with imaging evidence of progression free status lasting for at least 4 weeks after treatment, and without hormone or antiepileptic treatment for at least 4 weeks;
7. Subjects with body cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) that need local treatment or repeated drainage, and which are poorly controlled by the investigators' judgment;
8. Concurrent other malignant tumors (except history of the following tumors that occurred and were cured 5 years ago: non-melanoma, skin cancer, carcinoma in situ or non-invasive tumor);
9. Clinically significant cardiac disease within 6 months before administration of the study drug, including: myocardial infarction, unstable angina pectoris, cerebrovascular accident or other acute and uncontrollable heart diseases; A history of clinically significant ventricular arrhythmias (such as persistent ventricular tachycardia, ventricular fibrillation, torsade de pointe ventricular tachycardia); New York Heart Association (NYHA) grade III or IV congestive heart failure; QTc > 470 ms (female) or > 450 ms (male) or Personal or family history of congenital long QT syndrome (Naring A, 2012); Arrhythmias requiring antiarrhythmic drug treatment (subjects with heart rate controllable atrial fibrillation > 1 month before the first administration of the study drug were eligible for inclusion);
10. Subjects with evidence of risk of gastric bleeding or gastric perforation are not suitable for inclusion according to the judgment of investigators;
11. Active colitis, including infectious colitis, radiation colitis and ischemic colitis, within 4 weeks before administration of the study drug;
12. Pyloric obstruction or persistent recurrent vomiting (defined as vomiting ≥ 3 times in 24 hours);
13. Peripheral neuropathy ≥ grade 2 (refer to NCI CTCAE 5.0);
14. Subjects with active hepatitis B or C (HBsAg positive and/or HBcAb positive with HBV DNA titer more than 1000 copies/mL or 200 IU/mL; HCV Ab positive with HCV RNA titer higher than the upper limit of normal value);
15. HIV positive or syphilis infection requiring systematic treatment;
16. Subjects who have received systemic immunosuppressive therapy, including glucocorticoids, within 2 weeks before administration of the study drug; Subjects allowed to use physiological replacement dose of hydrocortisone or similar drugs;
17. Subjects with active autoimmune diseases requiring systemic immunosuppressive therapy in the past 2 years;
18. Subjects received other clinical trial drugs within 28 weeks before administration of the study drug;
19. Subjects have received antibody conjugated drugs targeting CLDN 18.2 in the past;
20. Subjects who are not appropriate for this clinical trial at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 21 days after the first dose of SYSA1801
  DLT was defined as ≥grade 3 adverse events (per protocal and NCI CTCAE 5.0)related to the study drug that occurred in the first administration cycle (21 days) of SYSA1801
Recommended Phase 2 Dose (RP2D) | Up to 24 months(end of treatment)
  RP2D may be selected based on the Maximum tolerated dose(MTD), pharmacokinetic and antitumor activity data
Incidence, severity, and outcome of adverse events (AEs) and serious adverse events (SAEs) | Up to 30 days after the last dose of SYSA1801
  The adverse events occurring or worsening on or after the first dose of the study drug will be recorded

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Predose and multiple timepoints up to 21 days after every dose (stage I)
  Cmax of SYSA1801, total antibodies and free MMAE
Time to maximum concentration(Tmax) | Predose and multiple timepoints up to 21 days after every dose (stage I)
  Tmax of SYSA1801, total antibodies and free MMAE
Area under the plasma concentration versus time curve (AUC) | Predose and multiple timepoints up to 21 days after every dose (stage I)
  AUC of SYSA1801, total antibodies and free MMAE
Immunogenicity: anti-drug antibody(ADA) | Predose and multiple timepoints up to 21 days after every dose (stage I)
  Antibodies against SYSA1801, including neutralizing antibodies
Objective Response Rate (ORR) | Up to 24 months(end of treatment)
  ORR was defined as the proportion of patients achieving either a confirmed complete response or partial response (PR), per RECIST v1.1
Disease Control Rate (DCR) | Up to 24 months(end of treatment)
  DCR is the proportion of patients with disease control (include patients with Complete response, partial response and stable disease)
Progression Free Survival (PFS) | Up to 24 months(end of treatment)
  PFS is defined as the time from the date of first administration to the date of the first documentation of progressive disease or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, Ph.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China